CLINICAL TRIAL: NCT06798610
Title: The Impact of the Inflammation Index on Predicting Postoperative Complications in Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, OSMAN KÖSE, MD, assistant professor, Sakarya University
Other Study IDs: E.309436-346
Record Dates: First submitted 2025-01-15; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Complications; Ovarian Cancer
Keywords: inflammation markers; complications; ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent cytoreductive surgery due to advanced-stage ovarian cancer: The study will investigate the complications that develop within one month following cytoreductive surgery in patients with advanced-stage ovarian cancer. It will explore the relationship between these complications and preoperative inflammatory markers

SUMMARY:
Advanced-stage ovarian cancer surgery is a procedure that inherently carries a high risk of mortality and morbidity. However, there are some uncertainties regarding whether these complications can be predicted before the operation. In this study, we aimed to examine the relationship between complications and inflammation.

DETAILED DESCRIPTION:
Objective: Cytoreductive surgery (CRS) is the most important treatment method that increases survival in advanced-stage ovarian cancer patients. However, complications after CRS are seen as a significant cause of morbidity and mortality. Preoperative risk assessment of patients is of great importance. In recent years, inflammatory markers have been the subject of many studies evaluating malignancy and surgical outcomes. Neutrophil-lymphocyte ratio (NLR), platelet-lymphocyte ratio (PLR), systemic inflammation index (SII), and systemic inflammatory response index (SIRI) stand out as prognostic and predictive tools in malignancies. This study aims to evaluate the preoperative inflammatory markers in patients who underwent CRS for advanced-stage epithelial ovarian cancer and to investigate the predictive power of postoperative complications.

Materials and Methods: This retrospective study examines patients who underwent CRS due to advanced-stage epithelial OC at Sakarya University Training and Research Hospital between 2014 and 2023. Postoperative complications of the patients were graded according to the Clavien-Dindo classification; NLR, PLR, SII, and SIRI values were calculated using preoperative laboratory data, and the predictive values of inflammatory markers were analyzed with ROC curves.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria of the patients were determined as those who underwent surgery with the diagnosis of FIGO Stage IIIc and IV epithelial ovarian cancer.

Exclusion Criteria:

* The exclusion criteria of the study were patients who had recently undergone blood transfusion or bacterial or viral infection within two weeks before surgery.
* Pregnant patients or patients with hematological diseases.
* Patients with thrombotic diseases.
* Patients with immunological diseases.
* Patients with severe liver or kidney diseases, patients with a previous history of cancer.
* Patients receiving anticoagulant and/or antiplatelet therapy due to venous or arterial thromboembolism.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study includes patients who underwent cytoreductive surgery for FIGO Stage IIIc and IV epithelial ovarian cancer between January 1, 2014, and December 31, 2023. Individuals who had received blood transfusion or had an infection prior to surgery, those with immunological or hematological diseases, patients with an ECOG performance score >3, those with a history of cancer, patients with venous thromboembolism history, and those recommended for neoadjuvant chemotherapy were excluded. Participants were evaluated for complications that could develop within 30 days after surgery.
Sampling Method: Non-Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Correlation Between Preoperative Inflammatory Markers and Postoperative Complications | Preoperative inflammatory markers will be measured within 1 week before surgery. Postoperative complications will be assessed within 30 days after surgery.
  This measure will examine the relationship between preoperative inflammatory markers and postoperative complications. The levels of inflammatory markers may be used to predict the risk of complications and can guide treatment approaches aimed at improving the recovery process following surgery.

CONTACTS AND LOCATIONS:
Overall Officials: osman köse, ass. proff., Study Director — Sakarya University Faculty of Medicine
Locations (2):
- Turkey (Türkiye) (2):
  - Sakarya University Faculty of Medicine, Adapazarı, Sakarya
  - Sakarya University Faculty of Medicine, Sakarya

IPD SHARING:
Plan to Share IPD: No